CLINICAL TRIAL: NCT06525155
Title: Effect of GnRH Agonist Administration on Decreasing VAS, Estradiol, and Anti Mullerian Hormone in Endometriosis Cyst Patients
Brief Title: Effect GnRH Agonist Administration in Endometriosis Cyst Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, Surya Adi Pramono, Principal Investigator, Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMR0123
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis
Keywords: Triptorelin embonate; Endometriosis cyst
MeSH Terms: conditions — Endometriosis | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Experimental): Triptorelin Embonate, 3 times dosing
  Interventions: Drug: Triptorelin Embonate
- Treatment 2 (Experimental): Triptorelin Embonate, 1 time dosing
  Interventions: Drug: Triptorelin Embonate

INTERVENTIONS:
Drug: Triptorelin Embonate — Treatment 1: 3.75 mg twice before surgery (baseline and week-6) and once after surgery at week-12
  Other Names: Pamorelin
  Arms: Treatment 1
Drug: Triptorelin Embonate — Treatment 2: 3.75 mg once after surgery at week-12
  Other Names: Pamorelin
  Arms: Treatment 2

SUMMARY:
Endometriosis is a chronic disease that affects 10-15% of women of childbearing age. The most common symptom is pelvic pain. One of the treatment options that has been proven effective in treating endometriosis symptoms, including endometriosis pain, is triptorelin. Triptorelin has also received a distribution permit in Indonesia for the treatment of endometriosis.

However, patient compliance in using this drug is very low due to high medical costs and side effects of the drug. Standard treatment with triptorelin is generally given every 4 weeks. A previous preliminary study showed that triptorelin could be given at 6-week interval and provided treatment results that were no different from those at 4-week interval. This is certainly better, because with longer interval doses it can reduce medical costs, reduce side effects due to hormone suppression and can increase patient compliance in undergoing treatment. Therefore, in this study triptorelin will be given to 2 groups and observed for 18 weeks. The first group will be given triptorelin twice before surgery, each with an interval of 6 weeks, at baseline and week-6. Then triptorelin will be given again once after surgery at week-12. In the second group, triptorelin will be given once after surgery at week-12. In this study, the effect of triptorelin on the treatment of endometriosis will be measured based on the improvement in the degree of pain felt by the subjects using a visual analogue scale (VAS) at baseline, week-6, week-12 (prior to surgery) and week-18; Anti Mullerian Hormone (AMH) levels, and estradiol levels before triptorelin administration (at baseline) and prior to surgery (week-12). The condition of the uterus and cysts will also be evaluated at the time of surgery.

DETAILED DESCRIPTION:
There will be 2 groups of treatment; each group will consist of 16 subjects with study period for 18 weeks.

Treatment I : twice before surgery (baseline and week-6) and once after surgery at week-12 Treatment II : once after surgery at week-12

The eligible subjects will be allocated to receive study medication (Treatment 1 or Treatment 2) in an open label study. They will be asked to come to the hospital every 6-week interval throughout the study period.

Subjects will be evaluated based on the improvement in the degree of pain felt by the subjects using a visual analogue scale (VAS) on each visit throughout the study period (at baseline, week-6, week-12 prior to surgery and week-18), and Anti Mullerian Hormone (AMH) levels and estradiol levels at baseline and week-12 (prior to surgery). The condition of the uterus and cysts will also be evaluated at the time of surgery at week-12.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18 to 40 years.
* The subjects was diagnosed with endometriosis cysts.
* Willing to participate in research and sign informed consent before all research-related activities begin.
* Regular menstruation (within 25 - 35 day intervals) in the last 3 months before the study was conducted.

Exclusion Criteria:

* The patient used hormonal contraception in the last 3 months prior to the study.
* Using a GnRH agonist within the past 3 months.
* Using the hormone progesterone within the last 3 months
* Pregnancy, breastfeeding females
* History of osteoporosis
* History of blood clotting disorders
* History of heart and blood vessel disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Anti Mullerian Hormones (AMH) levels | Baseline, week-12 (prior to surgery)
  Hormone which is produced by ovarian follicles indirectly represent remaining ovarian reserves.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline, week-6, week-12, week-18
  Pain intensity measurement tool and presented in the form of a horizontal line and given a number 0-10.
Estradiol levels | Baseline, week-12 (prior to surgery)
  Estradiol is a sex hormone that has proinflammatory and anti-apoptotic effects on endometrial cells which can exacerbate endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Surya A Pramono, Sp.OG., Subsp.FER, MD, Principal Investigator — Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Locations (1):
- Department of Obstetrics and Gynecology Central Army Hospital Gatot Soebroto, Jakarta, Indonesia